CLINICAL TRIAL: NCT00275704
Title: Phase II Evaluation of Flaxseed for the Treatment of Hot Flashes
Brief Title: Flaxseed for the Treatment of Hot Flashes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sandhya Pruthi, M.D., Mayo Clinic Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC04C9; MC04C9 (Other: Mayo Clinic Cancer Center); 247-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Linseed Oil

INTERVENTIONS:
Drug: Flaxseed

SUMMARY:
Flaxseed, a phytoestrogen, is a natural food supplement rich in plant ligands, which have a very weak estrogen effect. In this study, flaxseed is being evaluated in regard to its capacity to safely and effectively treat hot flashes. Specifically, this study seeks to determine if flaxseed will lower the number and severity of hot flashes and if women experience any side effects from taking flaxseed for this purpose.

ELIGIBILITY:
Inclusionary Criteria:

* Age greater than or equal to 18 years
* Women with a history of breast cancer (currently without malignant disease) or women who have no history of breast cancer but who wish to avoid estrogen due to a perceived increased risk of breast cancer.
* Bothersome hot flashes (defined by occurenece of greater than or equal to 14 times per week and of sufficient severity to make the patient desire therapeutic intervention).
* Presence of hot flashes for greater than or equal to 1 month prior to study entry.
* Life expectancy greater than or equal to 6 months.
* ECOG Performance Status (PS) 0 or 1 (see Appendix VIII)

Exclusionary Criteria/Contraindications

* Any of the following current (less than or equal to 4 weeks) or planned therapies (tamoxifen, raloxifene, or aromatase inhibitors are allowed, but patient must have been on a constant dose for greater than or equal to 4 weeks and must not be expected to stop the medication during the study period): antineoplastic chemotherapy, androgens, estrogens, progestational agents, other herbal supplements, including soy (herbal teas from a grocery store are allowed), warfarin (1 mg of daily warfarin is allowed for central line patency)
* History of allergic or other adverse reaction to flaxseed, wheat, nuts, lactose, and/or certain spices
* Current or planned use of other agents for treating hot flashes (except stable dose of vitamine E or antidepressants are allowed as long as they wre started >30 days prior to study initiation and are to be continued through the study period).
* Diabetes (as flaxseed can lower blood glucose levels and might have additive effects when used with antidiabetic drugs).
* Diagnosis of/problems with chronic diarrhea or history of bowel obstruction or esophageal stricture.
* Any of the following: pregnant women, nursing women, women of childbearing potential who are unwilling to employ adequate contraception
* Current use of anticoagulants including aspirin, clopidogrel (Plavix), ticlopidine (Ticlic), and coumadin (1 mg of dialy coumadin is allowed for central line patency).
* Diagnosis of/problems with von Willebrand's disease or other bleeding disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-05; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Determine if flaxseed will lower the number and severity of hot flashes
Determine if there are any side effects from taking flaxseed for hot flashes
Evaluate the impact of flaxseed on hot flash scores in women with a history of breast cancer or women who do not wish to take estrogen therapy for fear of increased risk of breast cancer.
Evaluate the toxicity of flaxseed in this study population.
Evaluate the effect of flaxseed on quality-of-life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Pruthi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States